CLINICAL TRIAL: NCT04782336
Title: Sample Collection to Facilitate the Performance Evaluation of the LumiraDx Point of Care Device for the Detection of Influenza A/B, Respiratory Syncytial Virus (RSV) & COVID-19 (SARS-COV-2 Virus)
Brief Title: Sample Collection Study to Aid Evaluation of an Influenza A/B, Respiratory Syncytial Virus & COVID-19 Virus POC Test
Acronym: INFORM
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment Pause
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00018
Record Dates: First submitted 2021-02-17; First posted 2021-03-04 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Covid19; RSV Infection; Influenza Type A; Influenza Type B
Keywords: POC; SARS-CoV-2; Antigen; Paediatric; Flu
MeSH Terms: conditions — COVID-19; Respiratory Syncytial Virus Infections; Influenza, Human | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sample Collection - Symptomatic Patients (Other): The patient will be completing or has completed a SOC Influenza A/B and/or COVID-19 and/or RSV test on the day of study
  Interventions: Other: Sample Collection

INTERVENTIONS:
Other: Sample Collection — Sample Collection - Adult Population:
  * Two (2) Nasal AND/OR
  * Two (2) Throat Swabs AND/OR
  * One (1) Saliva Sample
  Sample Collection - Paediatric Population:
  * Two (2) Nasal OR
  * Two (2) Throat Swabs AND/OR
  * One (1) Saliva Sample

SUMMARY:
Collection of Nasal Swabs, Throat Swabs and Saliva Samples from patients presenting at their designated care or testing facility displaying symptoms of either Influenza, Respiratory Syncytial Virus (RSV), SARS-CoV-2 or those who have been in recent contact with SARS-CoV-2 positive patients. Collected samples will aid the development, calibration and performance evaluation of the LumiraDx POC Test.

DETAILED DESCRIPTION:
INFORM is a sample collection study targeting a population of patients attending their designated care or testing facility, suspected of having a respiratory illness typical of Influenza, RSV or COVID-19 and undergoing a Standard of Care (SOC) test on the day. Or those who have been in recent contact with SARS-CoV-2 positive patients. Participants may be of any age, there is no upper or lower age limit.

Depending on the facility's viability and agreed contracting, the following study samples will be collected per patient:

Adult Population: Two (2) Nasal, AND/OR Two (2) Throat Swabs AND/OR, One (1) Saliva Sample

Paediatric Population: Two (2) Nasal, OR Two (2) Throat Swabs AND/OR, One (1) Saliva Sample

Once required samples and data have been collected, participation is complete. No follow-up or subsequent patient involvement is required.

ELIGIBILITY:
Inclusion Criteria:

* Preliminary assessment of the patient by the Investigator/Designee should be suggestive of Influenza and/or COVID-19 and/or RSV at the time of the study visit. This may include referral to a testing facility.
* The patient will be completing or has completed a Standard of Care (SOC) Influenza A/B, COVID-19 and/or an RSV test on the day of study. This SOC sampling can be conducted prior or post the patient consenting to this study.
* Written Informed Consent must be obtained prior to study enrolment:

  * A participant who is 16 years or older must be willing to give written informed consent and must agree to comply with study procedures.
  * The Legal Guardian or Legal Authorised Representative of a participant who is under the age of 16 must give written informed consent and agree to comply with study procedures. Active written assent should be obtained from children of appropriate intellectual age (as determined by the consent taker in accordance with GCP).

Exclusion Criteria:

* The patient underwent a nasal wash/aspirate as part of standard of care testing during their current visit.
* The patient is undergoing treatment currently and/or within the past 14 days of the study visit with an inhaled influenza vaccine (FluMist®) or anti-viral medication, which may include but is not limited to Amantadine (Symmetrel®), Rimantadine (Flumadine®), Zanamivir (Relenza®), Oseltamivir (Tamiflu®), or Baloxavir Marboxil (Xofluza™).
* The patient is undergoing treatment currently or had undergone within the past 14 days of the study visit with RSV-related medication which may include but is not limited to Ribavirin (Virazole), RSV-IGIV (RespiGam) or palivizumab (Synagis).
* The patient is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
* The patient does not have the capacity to consent as determined by the Research Team.
* The patient is deemed to be unsuitable for research at the Research Team's discretion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Collection of Nasal Swabs, Throat Swabs and Saliva Samples across a range of demographics. | 1-3 Years
  The collection of Nasal Swabs, Throat Swabs and Saliva Samples positive for Influenza A, Influenza B, RSV or SARS-CoV-2 across a range of demographics to help determine the accuracy of the LumiraDx Point of Care (POC) Influenza A/B + RSV and SARS-CoV-2 tests.

CONTACTS AND LOCATIONS:
Overall Officials: Samer Elkhodair, Principal Investigator — University College London Hospitals
Locations (6):
- United Kingdom (6):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - NHS Lothian - Royal Hospital for Children & Young People, Edinburgh
  - Leicester Royal Infirmary, Leicester
  - Barts Health NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation, London